CLINICAL TRIAL: NCT06983834
Title: The Effect of Mindfullness-Based Psychoeducation Applied to Primary Caregivers of Individuals With Bipolar Disorder on Caregivers' Mindfulness, Care Burden, Quality of Life and Psychological Resilience
Brief Title: Mindfulness Psychoeducation for Bipolar Disorder Caregivers' Mindfulness, Burden, Quality of Life and Resilience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Azime Korkmaz, PhD student, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PAU-SBE-AK-01
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: The study included two groups: an experimental group and a control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregivers of Bipolar Disorder Patients (Experimental) (Experimental): Mindfulness-based psychoeducation will be applied to the experimental group.There will be pre-test and post-tests.
  Interventions: Behavioral: Psychoeducation
- Caregivers of Bipolar Disorder Patients (Control) (No Intervention): Only pre-test and post-tests will be applied without any intervention.

INTERVENTIONS:
Behavioral: Psychoeducation — Mindfulness Based Psychoeducation
  Arms: Caregivers of Bipolar Disorder Patients (Experimental)

SUMMARY:
This study was designed to determine the effect of mindfulness-based psychoeducation applied to primary caregivers of individuals diagnosed with bipolar disorder on their mindfulness, caregiver burden, quality of life, and psychological resilience.

DETAILED DESCRIPTION:
Bipolar disorder is a chronic mental illness characterized by alternating episodes of opposing mood states (mania/hypomania and depression) and euthymic periods. Providing continuous care to individuals diagnosed with bipolar disorder can be highly challenging. Considering factors such as medication management, hospital follow-ups, patient behavior during episodes, and their attitudes toward themselves and others, being a primary caregiver is a demanding responsibility. Caregivers may face challenges such as constant caregiving burden, social isolation, burnout, neglecting self-care, and ignoring their own need for help. However, due to their perceived obligation to prioritize the patient, they may find themselves without adequate support.

Psychiatric nurses should approach not only the chronically mentally ill patient but also their caregivers, who are integral parts of the patient's environment, from a holistic perspective. The home environment of the patient, and particularly the attitude of the family and primary caregiver, plays a significant role in the prevention of relapses. From this holistic point of view, psychoeducation programs are expected to increase caregivers' psychological resilience, quality of life, and mindfulness levels, while reducing their caregiving burden. Such outcomes are anticipated to not only benefit the caregiver and the patient but also strengthen the broader society, as they may contribute to the reduction of relapse rates. Consequently, this could positively impact the national economy by decreasing healthcare utilization. Protecting caregivers may also lead to a reduced need for healthcare services directed toward them.

Psychoeducation is one of the core roles of psychiatric nurses. The recognition and expansion of mindfulness-based psychoeducation practices in the field are expected to provide significant support to both patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older,
* At least a primary school graduate,
* Able to hear, understand spoken language, and communicate,
* Has been a primary caregiver for at least 6 months and is participating voluntarily.

Exclusion Criteria:

* Currently participating in another psychoeducation group,
* Diagnosed with any mental disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
The Descriptive Characteristics Form | 6 months
  The Descriptive Characteristics Form consists of 16 questions related to individuals' sociodemographic information and personal characteristics (Age, Gender, Marital Status, Educational Status, Employment Status, Income Level, Caregiving Support, Duration of Being the Primary Caregiver, Smoking and Alcohol Use, Hobby Status, Social Support Information). It is a data collection tool developed based on a literature review.

SECONDARY OUTCOMES:
Zarit Burden Interview | 6 months
  The scale was developed by Zarit, Reever, and Bach-Peterson to measure caregiver burden.It is a scale that can be completed either by the caregivers themselves or through interviews conducted by the researcher. The scale uses a Likert-type rating system ranging from 0 to 4 (never, rarely, sometimes, quite frequently, nearly always). Scores on the scale range from 0 to 88. The items primarily focus on social and emotional aspects, and a higher total score indicates a greater level of burden or distress experienced by the caregiver.
The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36, Short Form-36 Health Survey) | 6 months
  The SF-36 Survey was developed by Ware and Sherbourne (1992) to assess quality of life.This scale is used to assess physical and mental health in individuals over the age of 14, whether they have various health conditions or are healthy. The SF-36 is a generic quality of life scale and provides a comprehensive evaluation. The scale consists of 36 items, which include: physical functioning (10 items), role limitations due to physical health problems (2 items), social functioning (2 items), role limitations due to emotional problems (3 items), mental health (5 items), vitality (4 items), bodily pain (2 items), general health perceptions (5 items), and perceived change in health status (1 item). Each item is evaluated individually and scored on a scale from 0 to 100.
Resilience Scale for Adults | 6 months
  The scale was developed by Friborg et al. (2003) to measure psychological resilience in adults. The scale consists of 33 items and 6 subscales: self-perception, perception of the future, structured style, social competence, family cohesion, and social resources. It is a 5-point Likert-type scale. The response options are scored as follows: 1 - Strongly Disagree, 2 - Disagree, 3 - Neutral, 4 - Agree, and 5 - Strongly Agree.
Mindful Attention Awareness Scale | 6 months
  The scale was developed by Brown and Ryan (2003) to measure the level of mindfulness and consists of 15 items.In the scale, each item is scored based on how frequently the individual experiences that specific situation. It is a 6-point Likert-type scale with the following response options: "Almost never: 6," "Very rarely: 5," "Rarely: 4," "Sometimes: 3," "Often: 2," and "Almost always: 1." The total score on the scale ranges from a minimum of 15 to a maximum of 90. Based on the total score, individuals scoring between 66 and 90 are considered to have a high level of mindfulness, scores between 41 and 65 indicate a moderate level, and scores of 40 or below reflect a low level of mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay TAŞDEMİR, AssocProfDr, Study Director — https://akbis.pau.edu.tr/personel/226
Locations (1):
- Afyonkarahisar University of Health Sciences, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No